CLINICAL TRIAL: NCT02961374
Title: Phase II Trial of Weekly Erlotinib Dosing to Reduce Duodenal Polyp Burden Associated With Familial Adenomatous Polyposis
Brief Title: Erlotinib Hydrochloride in Reducing Duodenal Polyp Burden in Patients With Familial Adenomatous Polyposis at Risk of Developing Colon Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2016-01674; NCI-2016-01674 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); N01-CN-2012-00042; MAY2016-07-01 (Other: Mayo Clinic in Rochester); MAY2016-07-01 (Other: DCP); N01CN00042 (NIH); P30CA015083 (NIH)
Record Dates: First submitted 2016-11-10; First posted 2016-11-11 (Estimated); Results first posted 2021-09-22 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Attenuated Familial Adenomatous Polyposis; Familial Adenomatous Polyposis
MeSH Terms: conditions — Attenuated familial adenomatous polyposis; Adenomatous Polyposis Coli | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (erlotinib hydrochloride) (Experimental): Patients receive erlotinib hydrochloride PO once weekly. Treatment continues for up to 6 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Erlotinib; Drug: Erlotinib Hydrochloride

INTERVENTIONS:
Drug: Erlotinib — Given PO
Drug: Erlotinib Hydrochloride — Given PO
  Other Names: Cp-358,774; OSI-774; Tarceva

SUMMARY:
This phase II trial studies the side effects of erlotinib hydrochloride and how well it works in reducing duodenal polyp burden in patients with familial adenomatous polyposis at risk of developing colon cancer. Erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the mean percent change in duodenal polyp burden (sum of diameters from all polyps) from baseline to 6 months post-intervention for familial adenomatous polyposis (FAP) subjects receiving weekly erlotinib hydrochloride (erlotinib).

II. To assess the grade 2/3 adverse event rate in this population and compare it to historical data.

SECONDARY OBJECTIVES:

I. To evaluate all adverse events at least possibly attributed to weekly erlotinib.

II. To assess the absolute and percent change in duodenal polyp number from baseline to 6 months.

III. To assess the absolute and percent changes in lower gastrointestinal polyp burden and number for the subset of participants with ileal pouch anal anastomosis (IPAA) or ileo-rectal anastomosis with rectal stump.

IV. To assess the absolute and percent change in desmoid tumor size in participants who have baseline and follow up computed tomography (CT)s performed as part of their standard of care.

CORRELATIVE OBJECTIVES:

I. Gene expression profiles in duodenal adenomas and uninvolved tissue will be compared between baseline and endpoint samples using negative binomial statistics (DESeq2).

II. Identify differentially expressed genes between duodenal polyps and uninvolved tissue at endpoint compared to baseline.

III. Evaluate the effect of weekly erlotinib on EGFR and Wnt target gene expression in duodenal adenomas.

IV. Evaluate the effect of weekly erlotinib on immune response signaling in duodenal adenomas and uninvolved tissue.

OUTLINE:

Patients receive erlotinib hydrochloride orally (PO) once weekly. Treatment continues for up to 6 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION INCLUSION
* Diagnosis of familial adenomatous polyposis (FAP) or attenuated familial adenomatous polyposis (AFAP), defined as at least one of the following:

  * Genetic diagnosis with confirmed APC mutation (Clinical Laboratory Improvement Act [CLIA] certified lab or research testing)
  * Obligate carrier
  * Clinical diagnosis of classic FAP with >= 100 colorectal adenomas status post colectomy and a family history of FAP
  * Clinical diagnosis of FAP, based on personal and family history; Note: This criterion requires documented review and agreement from either the study chair or the Cancer Prevention Network (CPN) lead investigator
* Ability to understand and the willingness to sign a written informed consent document
* Willing to discontinue taking nonsteroidal anti-inflammatory drugs (NSAIDS) for 30 days prior to initiation of and during intervention; exception: use of =< 81 mg daily or =< 650 mg weekly aspirin is allowed
* Willing to discontinue smoking for the duration of study intervention
* Willing to provide mandatory biospecimens as specified in the protocol
* REGISTRATION INCLUSION
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Leukocytes (white blood cells [WBC]) >= 3,000/uL (>= 2,500/uL for African-American participants)
* Platelet count >= 100 x 10^9/L
* Hemoglobin >= 11.5 g/dL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Alkaline phosphatase =< 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) =< 2 x institutional upper limit of normal (ULN)
* Alanine aminotransferase (ALT)/serum glutamate pyruvate transaminase (SGPT) =< 2 x institutional upper limit of normal (ULN)
* Creatinine =< institutional upper limits of normal (ULN)
* Urinary testing results within institutional limits of normal or deemed clinically insignificant
* Spigelman 2-3
* Not pregnant or breast feeding; Note: the effects of erlotinib (Tarceva ) on the developing human fetus at the recommended therapeutic dose are unknown; for this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately; breastfeeding should be discontinued if the mother is treated with erlotinib
* Willing to use adequate contraception to avoid pregnancy or impregnation until 2 weeks after discontinuing study agent

Exclusion Criteria:

* PRE-REGISTRATION EXCLUSION
* Any prior treatment with erlotinib or other agent whose primary mechanism of action is known to inhibit EGFR
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to erlotinib
* Use of potent CYP3A4 inhibitors, including but not limited to ketoconazole, atazanavir, clarithromycin, indinavir, itraconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, troleandomycin, voriconazole, and grapefruit or grapefruit juice
* Use of potent CYP3A4 inducers, including but not limited to rifampicin, rifabutin, rifapentine, phenytoin, carbamazepine, phenobarbital, and St. John's wort
* Use of any other investigational agents =< 12 weeks prior to pre-registration
* Uncontrolled intercurrent illness or recent surgical procedure that in the opinion of the investigative team would limit compliance with study requirements, including, but not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Myocardial infarction =< 6 months prior to intervention
  * Severely impaired lung function
  * Nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the treatment with study intervention
  * Diagnosed liver disease, such as cirrhosis, chronic active hepatitis, or chronic persistent hepatitis
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations
* History of invasive malignancy =< 3 years prior to pre-registration; exception: adequately treated carcinoma of the cervix, carcinoma in situ, or basal or squamous cell carcinomas of the skin
* Individuals on anticoagulation medications who cannot safely discontinue the medication for at least 48 hours prior to the study endoscopy, as determined by the study investigator and/or participant's primary healthcare provider
* History of any upper gastrointestinal (GI) surgery that does not permit access to or evaluation of a 10 cm segment of the duodenum that includes the duodenal bulb, i.e. Whipple procedure or similar
* REGISTRATION EXCLUSION
* Histologically-confirmed high grade dysplasia (HGD), cancer, or polyp burden that is not quantifiable
* Regular (>= 2 times per week) use of drugs that alter the pH of the gastrointestinal tract (GI) tract, such as proton pump inhibitors (PPI) and antacids; exceptions: individuals who use prescription PPIs and have approval from their primary health care provider to replace the PPI with an H2 receptor agonist, i.e. ranitidine, for the duration of the trial will be eligible
* Gastrointestinal bleeding; note that the presence of any symptoms (dyspnea, fatigue, angina, weakness, malaise, melena, hematochezia, hematemesis, anemia, abdominal pain) will require clinical assessment to rule out gastrointestinal bleeding

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2020-02-23 (Actual); Study Completion 2021-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Niloy J Samadder, Principal Investigator — Mayo Clinic
Locations (8):
- United States (7):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
- University of Puerto Rico, San Juan, Puerto Rico

REFERENCES:
- [Derived] Stone JK, Mehta NA, Singh H, El-Matary W, Bernstein CN. Endoscopic and chemopreventive management of familial adenomatous polyposis syndrome. Fam Cancer. 2023 Oct;22(4):413-422. doi: 10.1007/s10689-023-00334-3. Epub 2023 Apr 29. PMID 37119510
- [Derived] Samadder NJ, Foster N, McMurray RP, Burke CA, Stoffel E, Kanth P, Das R, Cruz-Correa M, Vilar E, Mankaney G, Buttar N, Thirumurthi S, Turgeon DK, Sossenheimer M, Westover M, Richmond E, Umar A, Della'Zanna G, Rodriguez LM, Szabo E, Zahrieh D, Limburg PJ. Phase II trial of weekly erlotinib dosing to reduce duodenal polyp burden associated with familial adenomatous polyposis. Gut. 2023 Feb;72(2):256-263. doi: 10.1136/gutjnl-2021-326532. Epub 2022 May 30. PMID 35636921

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Erlotinib Hydrochloride): Patients receive 350 mg erlotinib hydrochloride PO once weekly. Treatment continues for up to 6 months in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (Erlotinib Hydrochloride)
Started | 46
Completed | 42
Not Completed | 4
Not completed — Adverse Event | 4

BASELINE CHARACTERISTICS:
Population: All patients that registered for protocol treatment are included in this analysis.
Arm/Group | Treatment (Erlotinib Hydrochloride)
Number analyzed (Participants) | 46
Age, Continuous [Median (Full Range); unit: years] | 42 [18 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 40
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 43
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  Puerto Rico | 4
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change in Duodenal Polyp Burden
Description: Assessed by esophagogastroduodenoscopy, the mean percent change was calculated by subtracting the sum of diameters from all polyps at baseline from the sum of diameters of all polyps at 6 months, then dividing by the sum of diameters from all polyps at baseline and multiplying by 100.
Time Frame: Baseline to 6 months post-intervention
Population: Of the 46 patients registered, 42 patients began protocol treatment and were assessed at both baseline and at the 6 month timepoint.
Measure: Mean (95% Confidence Interval); unit: percent change in Duodenal Polyp Burden
Arm/Group | Treatment (Erlotinib Hydrochloride)
Number analyzed (Participants) | 42
percent change in Duodenal Polyp Burden | -29.6 [-39.6 to -19.7]

2. Primary Outcome: Number of Participants With Grade 2/3 Adverse Event (AE)
Description: Assessed according to National Cancer Institute's (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. The number of patients reporting a grade 2 or higher event are reported.
Time Frame: Up to 7 months from registration
Population: All patients that registered and completed one course of treatment are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Erlotinib Hydrochloride)
Number analyzed (Participants) | 46
Participants | 33

3. Secondary Outcome: Number of Participants With Any Adverse Events
Description: Assessed according to NCI CTCAE version 4.0. All registered and treated participants will be evaluable for AEs from the time of their first dose of weekly erlotinib treatment. To evaluate the AE profile for this treatment, the maximum grade for each type of adverse event will be recorded for each participant and frequency tables will be reviewed to determine the overall patterns. The number of patients reporting a grade 1 or higher adverse event at least possibly related to treatment are reported.
Time Frame: Up to 7 months from registration
Population: All registered patients that began protocol treatment and were assessed for adverse events are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Erlotinib Hydrochloride)
Number analyzed (Participants) | 46
Participants | 41

4. Secondary Outcome: Change in Duodenal Polyp Number
Description: The number of duodenal polyps at baseline and the number of polyps remaining after 6 months of treatment will collected. The change in duodenal polyp number will be calculated for each patient by subtracting the baseline number of polyps from the 6 month number. Therefore a negative value indicates a decrease in the number of polyps present after 6 months. The median difference and standard deviation is reported.
Time Frame: Baseline to 6 months
Population: All patients that began protocol therapy and were assessed for duodenal polyp number at baseline and after 6 months are included in this analysis.
Measure: Median (Standard Deviation); unit: polyps
Arm/Group | Treatment (Erlotinib Hydrochloride)
Number analyzed (Participants) | 42
polyps | -12.8 (22.96)

5. Secondary Outcome: Absolute Change in Lower Gastrointestinal Polyp Burden
Description: Lower GI polyp burden was defined using the Pouch Exam form as either 1) the average diameter reported for pouch for participants with ileal pouch-anal anastomosis (IPAA), or 2) the average diameter reported for rectum for participants with ileorectal anastomosis (IRA) + rectal stump. Absolute change from baseline to month 6 are reported here.
Time Frame: Baseline to 6 months
Population: All registered participants who reported an average lower GI polyp diameter at both baseline and assessed at month 6 and were evaluable for change in lower GI polyp number.
Measure: Median (Inter-Quartile Range); unit: polyps
Arm/Group | Treatment (Erlotinib Hydrochloride)
Number analyzed (Participants) | 11
polyps | 0 [0 to 1]

6. Secondary Outcome: Percent Change in Lower Gastrointestinal Polyp Burden
Description: Lower GI polyp burden was defined using the Pouch Exam form as either 1) the average diameter reported for pouch for participants with ileal pouch-anal anastomosis (IPAA), or 2) the average diameter reported for rectum for participants with ileorectal anastomosis (IRA) + rectal stump. The percent change from baseline to month 6 are reported here.
Time Frame: Baseline to 6 months
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: Percent change in polyp burden
Arm/Group | Treatment (Erlotinib Hydrochloride)
Number analyzed (Participants) | 11
Percent change in polyp burden | 0 [0 to 25.0]

7. Secondary Outcome: Absolute Change in Lower Gastrointestinal Polyp Number
Description: Lower GI polyp number was defined using the Pouch Exam form as either 1) the number of polyps reported for pouch for participants with ileal pouch-anal anastomosis (IPAA), or 2) the number of polyps reported for rectum for participants with ileorectal anastomosis (IRA) + rectal stump. Absolute change from baseline to month 6 are reported here.
Time Frame: Baseline to 6 months
Population: All registered participants who reported total number of lower GI polyps at baseline and assessed at month 6 and were evaluable for change in lower GI polyp number.
Measure: Median (Inter-Quartile Range); unit: Change in the polyp number
Arm/Group | Treatment (Erlotinib Hydrochloride)
Number analyzed (Participants) | 18
Change in the polyp number | -6 [-26.0 to 0.0]

8. Secondary Outcome: Percent Change in Lower Gastrointestinal Polyp Number
Description: Lower GI polyp number was defined using the Pouch Exam form as either 1) the number of polyps reported for pouch for participants with IPAA, or 2) the number of polyps reported for rectum for participants with IRA + rectal stump.
Time Frame: Baseline to 6 months
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: percent change in polyp number
Arm/Group | Treatment (Erlotinib Hydrochloride)
Number analyzed (Participants) | 18
percent change in polyp number | -30.8 [-47.4 to 0.0]

9. Secondary Outcome: Absolute and Percent Change in Desmoid Tumor Size
Description: Laboratory measures will be correlated with participant outcomes (i.e., polyp burden, adverse events) and with each other as well. Cut-points will be determined based on previously defined and accepted standards. Descriptive statistics and simple scatter plots will be generated to review the tissue-based biomarker data. For continuous variables, the actual and % change in the level of each of the biomarkers from pre- to post-intervention will be explored using Wilcoxon signed rank tests, and paired sample t-tests. All categorical variables will be analyzed using chi-square tests or Fisher's exact test. For all translational endpoints, any notable statistical result will be viewed as an impetus for further study rather than as a definitive finding in and of itself.
Time Frame: Baseline to 6 months
Population: Data on desmoid tumor size was not collected.
Arm/Group | Treatment (Erlotinib Hydrochloride)
Number analyzed (Participants) | 0

10. Other Pre Specified Outcome: Immune Response Signaling in Duodenal Adenomas and Uninvolved Tissue
Description: as for outcome 9
Time Frame: Up to 2.5 years
Reporting Status: Not Posted

11. Other Pre Specified Outcome: EGFR and Wnt Gene Expression
Description: as for outcome 9
Time Frame: Up to 2.5 years
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Change in Differentially Expressed Genes of Duodenal Polyps and Uninvolved Tissue
Description: as for outcome 9
Time Frame: Baseline to 2.5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected monthly for up to 7 months from registration.
Description: Adverse events were collected monthly for up to 7 months from registration.
Arm/Group | Treatment (Erlotinib Hydrochloride)
All-Cause Mortality (participants affected / at risk) | 0/46
Serious Adverse Events (participants affected / at risk) | 3/46
Other Adverse Events (participants affected / at risk) | 46/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Erlotinib Hydrochloride) (N=46)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Reproductive system and breast -Oth spec (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Erlotinib Hydrochloride) (N=46)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Palpitations (Cardiac disorders) | 2 (3)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 2 (3)
Eye disorders - Other, specify (Eye disorders) | 1 (1)
Keratitis (Eye disorders) | 1 (1)
Photophobia (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (6)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 24 (47)
Dyspepsia (Gastrointestinal disorders) | 6 (6)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 3 (3)
Gastritis (Gastrointestinal disorders) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 3 (3)
Lip pain (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 3 (5)
Nausea (Gastrointestinal disorders) | 16 (22)
Oral pain (Gastrointestinal disorders) | 2 (2)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (9)
Fatigue (General disorders) | 12 (47)
Fever (General disorders) | 1 (1)
Flu like symptoms (General disorders) | 4 (4)
Gen disord and admin site conds-Oth spec (General disorders) | 4 (4)
Malaise (General disorders) | 4 (5)
Non-cardiac chest pain (General disorders) | 2 (2)
Pain (General disorders) | 2 (3)
Immune system disorders - Other, specify (Immune system disorders) | 2 (3)
Bronchial infection (Infections and infestations) | 2 (2)
Conjunctivitis (Infections and infestations) | 1 (2)
Enterocolitis infectious (Infections and infestations) | 2 (3)
Infections and infestations - Oth spec (Infections and infestations) | 3 (3)
Lip infection (Infections and infestations) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Rhinitis infective (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 3 (3)
Tooth infection (Infections and infestations) | 1 (3)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (3)
Vaginal infection (Infections and infestations) | 1 (1)
Prolapse of intestinal stoma (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 4 (7)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Metabolism, nutrition disord - Oth spec (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 7 (15)
Dysgeusia (Nervous system disorders) | 2 (2)
Dysphasia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 12 (29)
Paresthesia (Nervous system disorders) | 1 (2)
Syncope (Nervous system disorders) | 1 (1)
Vasovagal reaction (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3)
Irritability (Psychiatric disorders) | 1 (1)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (3)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1)
Dysmenorrhea (Reproductive system and breast disorders) | 1 (1)
Reproductive system and breast -Oth spec (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (7)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (6)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (6)
Rash acneiform (Skin and subcutaneous tissue disorders) | 25 (54)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 5 (8)
Hypertension (Vascular disorders) | 1 (4)
Superficial thrombophlebitis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-22): https://cdn.clinicaltrials.gov/large-docs/74/NCT02961374/Prot_SAP_000.pdf